CLINICAL TRIAL: NCT06292871
Title: The Acceptability and Feasibility of Using a Social Media Platform to Provide Continuous Support in the Follow-up Management of Gestational Diabetes: A Pilot Randomised Controlled Trial
Brief Title: The Use of Social Media Platform to Continuously Support Pregnant Women With Gestational Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singapore Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/2712
Record Dates: First submitted 2024-02-21; First posted 2024-03-05 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-02

CONDITIONS: Gestational Diabetes
Keywords: Maternal Behaviour; Mobile Health; Blood Glucose; Emotional Wellbeing; Engagement
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: The study will employ a randomized controlled trial design, with GDM patients from KKH randomly assigned to either the intervention or control group. Randomization will be conducted via the electronic randomization list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Pregnant women with GDM receiving additional support via social media platform continuously for 1 month, in addition to the usual care management.
  Interventions: Behavioral: Additional GDM management through social media; Behavioral: Usual care
- Control Group (Active Comparator): Pregnant women with GDM under usual care management.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Additional GDM management through social media — Usual care provided by a diabetes nurse educator and dietitian. Additional educational resources for dietary management care received, and for any queries to be addressed by dietitian via social media platform from baseline to one-month follow-up visit.
  Arms: Intervention Group
Behavioral: Usual care — Usual care provided by a diabetes nurse educator and dietitian.

SUMMARY:
To assess the efficacy of utilizing a social media platform for dietary and lifestyle management in improving acceptance and blood glucose control in patients with gestational diabetes mellitus (GDM), compared to the control group under usual care. Specifically,

i. To measure the participants' acceptability and satisfaction levels of receiving intervention through the social media platform.

ii. To measure the feasibility of using the social media platform to provide GDM support through participants' engagement levels and feedback questionnaire.

iii. To measure the efficacy of using the social media platform to manage emotional responses in women with GDM.

iv. To measure the efficacy of using the social media platform to optimize glycemic control in women with GDM.

DETAILED DESCRIPTION:
Engaging pregnant women with GDM in dietary management over the gestation has been challenging. This pilot trial aims to assess the efficacy of utilizing a social media platform for dietary and lifestyle management in improving acceptance and blood glucose control among patients with GDM, compared to a control group receiving usual care. The study will employ a randomized controlled trial design, with GDM patients from KK Women's and Children's Hospital (KKH) randomly assigned to either the usual care (control; n=40) or to additional support via a dedicated social media platform for a period of 1 month, where a moderator will be available to address patients' queries and share relevant educational resources (intervention; n=40). Outcome measures include acceptance, satisfaction, and engagement levels, emotional well-being as well as the percentage achievement of time-in-range glucose readings for GDM patients. The independent t-test will be used to compare the outcome measures between groups. The findings from this study will provide valuable insights into the feasibility and efficacy of incorporating digital platforms into routine dietary counselling practices for improved patient outcomes and enhanced management of GDM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with GDM as confirmed by the Oral Glucose Tolerance Test during pregnancy
* Age ≥ 21 and ≤ 45 years
* Attended first (baseline) session of GDM diet counselling session
* Able to read and comprehend English
* Have a digital device accessible to social media platform
* Have SingPass access
* Able to provide informed consent

Exclusion Criteria:

* With known Type 1 or Type 2 diabetes
* Have multiple pregnancy

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Acceptance levels | At the end of one month from baseline visit
  Assessed by a 5-point Likert-type scale, ranging from 1 (completely disagree) to 5 (completely agree). A higher score indicates a higher acceptance level.
Satisfaction levels | At the end of one month from baseline visit
  Assessed by a 5-point Likert-type scale, ranging from 1 (completely disagree) to 5 (completely agree). A higher score indicates a higher satisfaction level.

SECONDARY OUTCOMES:
Engagement levels | At the end of one month from baseline visit
  Assessed by frequency of interactions with the platform moderator and frequency of platform visits among women in the intervention group
Appropriateness levels | At the end of one month from baseline visit
  Assessed by a 5-point Likert-type scale, ranging from 1 (completely disagree) to 5 (completely agree). A higher score indicates a greater appropriateness level.
Feasibility levels | At the end of one month from baseline visit
  Assessed by a 5-point Likert-type scale, ranging from 1 (completely disagree) to 5 (completely agree). A higher score indicates a higher feasibility level.
Emotional wellbeing | At the end of one month from baseline visit
  Assessed by the Perceived Stress Scale on a 5-point Likert-type scale, ranging from 0 (never) to 4 (very often). A higher score indicates a higher perceived stress level.
Blood glucose levels | At the end of one month from baseline visit
  Assessed by finger prick tests, in mmol/L
Proportion of participants with optimal blood glucose control | At the end of one month from baseline visit
  Based on recommended pre-meal range of 4.4-5.5 mmol/L and 2h post-meal range of 5.5-6.6 mmol/L

OTHER OUTCOMES:
Confidence levels | At the end of one month from baseline visit
  Assessed by a 5-point Likert-type scale, ranging from 1 (completely disagree) to 5 (completely agree). A higher score indicates a higher confidence level.
Meal skipping | At the end of one month from baseline visit
  Assessed by frequency of breakfast, lunch and dinner skipping a week
Proportion of participants with cigarette smoking | At the end of one month from baseline visit
  Assessed by active and passive smoking exposure, yes/no
Proportion of participants with alcohol intake | At the end of one month from baseline visit
  Assessed by current alcohol consumption, yes/no
Gestational weight gain rate | Throughout intervention period until delivery timepoint
  Weight gain per week, in kg/week
Proportion of participants with inappropriate weight gain | Throughout intervention period until delivery timepoint
  Defined by Institution of Medicine guideline for gestational weight gain
Motivational levels | At the end of one month from baseline visit
  Assessed by a 5-point Likert-type scale, ranging from 1 (lowest) to 5 (highest).
Proportion of participants with induced labour | At birth
  Based on onset of labour, retrieved from medical records
Proportion of participants with caesarean delivery | At birth
  Based on mode of delivery, retrieved from medical records
Birth weight | At birth
  Retrieved from medical records, in gram
Birth length | At birth
  Retrieved from medical records, in cm
Head circumference | At birth
  Retrieved from medical records, in cm
Birth size-for-gestational age | At birth
  Defined by percentile values, adjusted for gestational age at birth and sex
Gestational length at birth | At birth
  Retrieved from medical records, in weeks
Proportion of participants with preterm delivery | At birth
  Defined by gestational weeks at birth <37 weeks
Neonatal apgar score | At birth
  Retrieved from medical records, ranging from 0 (lowest) to 10 (highest). The higher the better.
Proportion of participants delivering healthy live birth | At birth
  Retrieved from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Wee Meng Han, PhD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hewage S, Audimulam J, Sullivan E, Chi C, Yew TW, Yoong J. Barriers to Gestational Diabetes Management and Preferred Interventions for Women With Gestational Diabetes in Singapore: Mixed Methods Study. JMIR Form Res. 2020 Jun 30;4(6):e14486. doi: 10.2196/14486. PMID 32602845
- [Background] Leblalta B, Kebaili H, Sim R, Lee SWH. Digital health interventions for gestational diabetes mellitus: A systematic review and meta-analysis of randomised controlled trials. PLOS Digit Health. 2022 Feb 24;1(2):e0000015. doi: 10.1371/journal.pdig.0000015. eCollection 2022 Feb. PMID 36812531
- [Background] Nguyen CL, Pham NM, Binns CW, Duong DV, Lee AH. Prevalence of Gestational Diabetes Mellitus in Eastern and Southeastern Asia: A Systematic Review and Meta-Analysis. J Diabetes Res. 2018 Feb 20;2018:6536974. doi: 10.1155/2018/6536974. eCollection 2018. PMID 29675432
- [Background] Yew TW, Chi C, Chan SY, van Dam RM, Whitton C, Lim CS, Foong PS, Fransisca W, Teoh CL, Chen J, Ho-Lim ST, Lim SL, Ong KW, Ong PH, Tai BC, Tai ES. A Randomized Controlled Trial to Evaluate the Effects of a Smartphone Application-Based Lifestyle Coaching Program on Gestational Weight Gain, Glycemic Control, and Maternal and Neonatal Outcomes in Women With Gestational Diabetes Mellitus: The SMART-GDM Study. Diabetes Care. 2021 Feb;44(2):456-463. doi: 10.2337/dc20-1216. Epub 2020 Nov 12. PMID 33184151